CLINICAL TRIAL: NCT06304350
Title: A Single Arm, Single Center, Phase II Clinical Study of Pembrolizumab Combined With Preoperative Chemotherapy (Albumin Paclitaxel+Carboplatin) Neoadjuvant Therapy for Resectable Locally Advanced (Stage II/III) Esophageal Squamous Cell Carcinoma
Brief Title: Pembrolizumab Combined With Preoperative Chemotherapy (Albumin Paclitaxel+Carboplatin) Neoadjuvant Therapy for Resectable Locally Advanced (Stage II/III) Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tongji University (Other)
Responsible Party: Principal Investigator, Jiang Fan, Director of Department of Thoracic Surgery, Tongji University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGHDOT-24-20
Record Dates: First submitted 2024-02-21; First posted 2024-03-12 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Esophageal Cancer
Keywords: esophageal cancer；; Pembrolizumab；; Neoadjuvant therapy
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination of pembrolizumab and platinum containing dual drugs (Experimental): After 2 courses of treatment with pembrolizumab combined with platinum containing dual drugs (albumin paclitaxel+carboplatin), surgery was performed, and postoperative pembrolizumab immunomaintenance therapy continued
  Interventions: Drug: Combination of pembrolizumab and platinum containing dual drugs

INTERVENTIONS:
Drug: Combination of pembrolizumab and platinum containing dual drugs — After 2 courses of treatment with a combination of pembrolizumab and platinum containing dual drugs (albumin paclitaxel+carboplatin), surgery was performed and pembrolizumab immunomaintenance therapy continued after surgery

SUMMARY:
This study is a prospective, single center, open label, single arm clinical study. Select resectable locally advanced (cT3-4aN0M0, cT1-3N1-2M0, cII/III stage) esophageal cancer with pathological diagnosis of squamous cell carcinoma for inclusion, receive pembrolizumab combined with platinum containing dual drug (albumin paclitaxel+carboplatin) treatment for 2 courses, and undergo surgery. After surgery, continue pembrolizumab immunotherapy. Using pCR as the main endpoint of the study

DETAILED DESCRIPTION:
This study is a prospective, single center, open label, single arm Phase II clinical study. Patients with locally resectable advanced esophageal squamous cell carcinoma were selected for inclusion in the study, who received a 2-course neoadjuvant treatment with pembrolizumab combined with platinum containing dual drugs. After evaluation, surgery was performed. The efficacy and safety of pembrolizumab combined with chemotherapy neoadjuvant therapy for resectable locally advanced esophageal squamous cell carcinoma were observed, with pCR and MPR as the main research endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Baseline stage resectable cII/III esophageal squamous cell carcinoma (8th UICC TNM stage);
2. Failure to receive anti-tumor treatment for esophageal squamous cell carcinoma;
3. Age range from 18 to 75 years old;
4. There are no surgical contraindications in the preoperative evaluation of various organ functions;
5. The following laboratory tests confirm that the bone marrow, liver and kidney functions meet the requirements for participating in the study: hemoglobin ≥ 9.0g/L; White blood cell count 4.0-10 × 109/L; Neutrophil absolute value (ANC) ≥ 1.5 × 109/L; Platelet count ≥ 100 × 109/L; Total bilirubin ≤ 1.5 times the upper limit of normal value; ALT and AST ≤ 2.5 times the upper limit of normal values; The international standardized ratio of prothrombin time is ≤ 1.5 times the upper limit of normal values, and some prothrombin time is within the normal range; Creatinine ≤ 1.5 times the upper limit of normal value;
6. Patients who have not undergone chemotherapy, radiation therapy, or hormone therapy for malignant tumors, have no history of other malignant tumors, and do not include prostate cancer patients who have received hormone therapy and have obtained DFS for more than 5 years;
7. Expected to achieve R0 resection;
8. Physical state ECOG 0-1;
9. The subjects must understand and sign the informed consent form

Exclusion Criteria:

1. Individuals who have received previous treatment for esophageal cancer (surgery, radiotherapy, chemotherapy, immunotherapy, targeted therapy, etc.);
2. Not suitable for surgery or with surgical contraindications;
3. Have a history of other anti PD-L1/PD-1 treatments;
4. Individuals with immunodeficiency or long-term systemic steroid therapy, or those who have received any immunosuppressive therapy within 7 days prior to receiving the study drug;
5. Individuals with active autoimmune diseases requiring systemic treatment within 2 years;
6. Patients with poor control of heart disease
7. Pregnant or lactating female patients;
8. For patients with drug allergies in the protocol.

Exit criteria：

Withdrawal cases refer to subjects who have stopped continuing treatment in clinical research due to various reasons. Subjects who experience the following situations will withdraw from the investigational treatment:

1. The main indicators are missing, and more than half of the items that can be filled in CRF are missing;
2. The surgical procedure violates the plan;
3. Cases that are excluded due to adverse reactions are not evaluated for efficacy, but side effects should be included in the statistics;
4. According to the researcher's opinion, continuing to participate in the study will be harmful to their health;
5. Patients who fail to undergo non-surgical treatment due to various reasons, including malignant tumor progression, underlying disease progression, patient or their trustee requesting withdrawal, will be reported together;
6. Missing subjects. All subjects who withdrew from the study should record their reasons for withdrawal in the CRF and their medical records. According to the ITT principle, all withdrawn cases should undergo survival analysis and toxicity evaluation for the corresponding group.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-02-17 (Actual); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete remission (pCR) | in two weeks after the surgical resection
  Defined as the absence of any residual esophageal squamous cell carcinoma cells, including the primary lesion and lymph nodes

SECONDARY OUTCOMES:
Major pathological remission (MPR) | in two weeks after the surgical resection
  The primary pathological response (MPR) is defined as residual survival tumor during surgery ≤ 10%.
R0 resection rate | in two weeks after the surgical resection
Progression free survival (PFS) | receiving therapy，up to approximately 2years.
Total survival time (OS) | The time from the patient's randomization receiving therapy to death from any cause，up to approximately 2years
Safety (incidence of adverse drug reactions) | Randomly group patients to receive treatment for up to two years

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No